CLINICAL TRIAL: NCT02447328
Title: A Single Arm, Tolerability and Safety Phase IV Study of Fulvestrant(Faslodex® ) as 2nd Line and Later Therapy in Postmenopausal Women With Locally Advanced or Metastatic Breast Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: D6998L00004
Record Dates: First submitted 2015-05-04; First posted 2015-05-18 (Estimated); Results first posted 2018-03-22 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Locally Advanced or; Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm (Experimental): Faslodex treated in the study
  Interventions: Drug: Fulvestrant

INTERVENTIONS:
Drug: Fulvestrant — fulvestrant (Faslodex®) 500mg/month for about 6 months with an additional 500mg dose given 14 days after the initial dose injection.

SUMMARY:
This single-arm study aims to assess the safety and tolerability profile of Fulvestrant(Faslodex®) as 2nd line and later therapy in postmenopausal women with locally advanced or metastatic breast cancer. The primary objective is to evaluate the adverse events after Fulvestrant (Faslodex®) for about 6 months

DETAILED DESCRIPTION:
This study is a Phase 4, single-arm, safety and tolerability study of fulvestrant (Faslodex®) as 2nd line therapy in postmenopausal women with locally advanced or metastatic breast cancer.

All of enrolled patients in this study will be injected fulvestrant (Faslodex®). This study will be performed for about 3 years and approximately 100 patients(actual target will be 80 treated patients) will be enrolled in about 10 investigational sites.

After obtaining the written informed consent from the patients, the information of demographic and medical history will be collected and laboratory tests will be performed.

Patients who meet the inclusion/exclusion criteria will be injected the fulvestrant (Faslodex®) 500mg/month for about 6 months with an additional 500mg dose given 14 days after the initial dose injection. The information of adverse events will be collected after the 1st dose of IP injection. In case that the evaluation of tumor response might be performed in regular clinical practice, those data will also be collected as well. The quality of life will also be measured.

ELIGIBILITY:
Inclusion Criteria:

* Post menopausal status women
* Outpatient or inpatient with locally advanced or metastatic breast cancer who have failed with prior anti-estrogen therapy.
* Estrogen receptor positive
* Radiographic progression of disease after the prior therapy
* Patients who agree to participate in this study and sign the informed consent

Exclusion Criteria:

* Patients who are treated with fulvestrant
* Patients who are being treated with the other antitumor agents
* Pregnancy or lactating women
* History of hypersensitivity to any of included ingredients (eg. Castor oil)
* Patients who are considered not fit for the study by investigators
* Patients who have severe dysfunction of liver or kidney

Ages: 18 Years to 130 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2015-05-29 (Actual); Primary Completion 2016-05-06 (Actual); Study Completion 2020-09-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- South Korea (6):
  - Research Site, Cheongju-si
  - Research Site, Daegu
  - Research Site, Goyang-si
  - Research Site, Seogu
  - Research Site, Seongnam-si
  - Research Site, Seoul

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject enrolled: 29MAY2015 Last subject last visit: 06MAY2016
  This study was conducted from 29 May 2015 to 06 May 2016 and 85 subjects from 9 study centres participated.
Pre-assignment Details: 1. Visit 1 (Enrolment visit) Obtained ICF and Eligibility check
  2. Duration of treatment with Fulvestrant (Faslodex®):
     Study drug administered biweekly at first cycle. Afterward, Study drug administered monthly. (expected duration of treatment: 6 cycles)
  3. End of Study post dose follow-up visit after study drug discontinuation.
Groups:
- Single Arm: fulvestrant (Faslodex®)
Period: Overall Study
Arm/Group | Single Arm
Started | 83 (Enrolment 85 Screening Failure 2 starting study drug 83)
Completed | 82
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: In this study, a total of 85 subjects were enrolled, and 83 of them received study drug open labelled, single arm. The safety population included 81 subjects who met all of the inclusion/exclusion criteria, and 74 of them were included in the efficacy population.
Arm/Group | Single Arm
Number analyzed (Participants) | 81
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age | 56.6 (9.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Safety(Percentage of Participants With Adverse Events and/or Adverse Drug Reactions)
Description: Percentage of patients with AEs.
Time Frame: Adverse events were collected from treatment initiation to end of the study about 6 months for each patient.
Population: The safety population: All patients given at least one dose of the study treatment will be included. Data from this population will be used for the safety analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Single Arm
Number analyzed (Participants) | 81
Percentage of participants
  Adverse Events(AE) | 81.5 [71.3 to 89.3]
  ADR; based on current South Korea label. | 38.3 [27.7 to 49.7]
  Serious AE | 11.1 [5.2 to 20.1]
  Serious ADR | 0 [0 to 4.4]
  Unexpected AE | 71.6 [60.5 to 81.1]
  Unexpected ADR | 24.7 [15.8 to 35.5]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Single Arm
Serious Adverse Events (participants affected / at risk) | 9/81
Other Adverse Events (participants affected / at risk) | 66/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm (N=81)
CHOLANGITIS (Hepatobiliary disorders) | 1 (1)
contusion of brain (Injury, poisoning and procedural complications) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1)
Acute lymphocytic leukaemia (in remission) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Joint Dislocation (Injury, poisoning and procedural complications) | 1 (1)
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
pelvic pain (Reproductive system and breast disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm (N=81)
back pain (General disorders) | 9 (11)
Pain (General disorders) | 6 (6)
fatigue (General disorders) | 5 (5)
nausea (Gastrointestinal disorders) | 10 (12)
Constipation (Gastrointestinal disorders) | 7 (7)
Anorexia (Gastrointestinal disorders) | 6 (6)
Dyspepsia (Gastrointestinal disorders) | 5 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 10 (12)
arthralgia (Musculoskeletal and connective tissue disorders) | 6 (6)
headache (Nervous system disorders) | 7 (7)
dizziness (Nervous system disorders) | 9 (10)
upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (5)
pruritus (Skin and subcutaneous tissue disorders) | 5 (5)
rash (Skin and subcutaneous tissue disorders) | 5 (5)

LIMITATIONS AND CAVEATS:
less information in efficacy set.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
14.1 The Institution and the Principal Investigator shall be entitled to publish the results of, or make presentations related to, the Study, provided that any publications or presentations to be made within 2 years of completion of the Study shall require the Company's prior written consent.